CLINICAL TRIAL: NCT00980278
Title: Cell Therapy Using Autologous Bone Marrow Cells Expanded Ex Vivo and Delivered Using Tricalcium Phosphate
Brief Title: Bone Tissue Engineering Using Autologous Bone Repair Cell (BRC) Therapy for Sinus Floor Bone Augmentation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, William Giannobile, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00014299
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-11

CONDITIONS: Tooth Loss
Keywords: sinus lift; tooth extraction; dental implant
MeSH Terms: conditions — Tooth Loss | interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sinus lift plus dental implant (Active Comparator): Transalveolar sinus augmentation will be performed. After 4 months dental implants will be delivered only if primary stability can be achieved.
  Intervention (Procedure/Surgery): Sinus lift augmentation and dental implant transalveolar sinus augmentation will be performed. After 4 months, dental implants will be delivered only if primary stability can be achieved.
  Biological/Vaccine: N/A; only sinus augmentation and dental implant
  Interventions: Procedure: Sinus lift augmentation and dental implant
- sinus lift plus BRCs and dental implant (Experimental): transalveolar sinus augmentation will be performed. A unit dose of BRC (10 ml) will be mixed with a commercially available β-TCP (Cerasorb), which will be used as a carrier to deliver the cells.
  Intervention (Procedure/Surgery): Sinus lift augmentation and dental implant transalveolar sinus augmentation will be performed. After 4 months, dental implants will be delivered only if primary stability can be achieved.
  Biological/Vaccine: Aastrom BRCs, sinus augmentation, BRC application, dental implant
  Interventions: Biological: Aastrom BRCs

INTERVENTIONS:
Procedure: Sinus lift augmentation and dental implant — transalveolar sinus augmentation will be performed. After 4 months, dental implants will be delivered only if primary stability can be achieved.
  Arms: sinus lift plus dental implant
Biological: Aastrom BRCs — sinus augmentation, BRC application, dental implant
  Arms: sinus lift plus BRCs and dental implant

SUMMARY:
The purpose of this research is to determine if one's own bone marrow tissue can help regenerate (grow) bone in the area of the jaw where an implant will be placed. The name of the process is called Bone Repair Cell (BRC) Therapy. A sample of bone marrow tissue will be collected and sent to a laboratory where it will be processed to form more cells. These new cells will then be transplanted in the regenerative site or sinus floor augmentation site. The researchers are testing to see if these cells (BRC) will help form bone indicating. The research will also determine if the implant will be more stable in the area with new bone growth.

DETAILED DESCRIPTION:
The overall aim is to promote bone regeneration, using Aastrom's proprietary Adult Stem Cell Therapy (AST) developed collaboratively with the University of Michigan, to enable placement of dental implants in patients who lack adequate alveolar bone. This project addresses specifically the placement of dental implants following bone regenerative sinus floor augmentation. This novel therapy mitigates the risks of other therapies, providing additional benefits of adequate cell numbers for high quality bone regeneration, and has the potential to become the new standard of care. In Aastrom's patented manufacturing technology, iliac bone marrow aspirates are expanded ex-vivo to enrich for adult multipotent cells (Bone Repair Cells- BRC) capable of regenerating bone and blood vessels. BRC will then be mixed with bone matrix graft extender, beta-tricalcium phosphate (β-TCP), before their implantation into the regenerative site.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 20-70 yrs
* Gender: Male and female
* Systemically healthy: Physical status according to the American Society of Anesthesiologists (ASA) I or II
* Requiring sinus augmentation to allow dental implant placement
* Missing teeth: Maxillary second premolar, maxillary first molar and/or maxillary second molar
* Remaining alveolar bone height: 2 to 6 mm
* Must be able and willing to follow study procedures and instructions
* Must have read, understood and signed an informed consent form

Exclusion Criteria:

* Allergies or hypersensitivities to study related medications: dexamethasone, chlorhexidine, ibuprofen. For patients allergic to amoxicillin a comparable substitute antibiotic will be used
* Hematologic disorders/ blood dyscrasias
* Active infectious disease
* Liver or kidney dysfunction/failure- Patients will have blood drawn for serum laboratory tests, including creatinine, blood urea nitrogen, AST, ALT, and bilirubin. All of these must be within normal limits for a patient to be included in the study
* Laboratory values that will define normal renal and hepatic function, as well as criteria for exclusion of metabolic bone disease are consistent with those established by the University of Michigan Health System (UMHS). Normal clinical values will be used to help assure the health of all subjects in this trial. Potential subjects whose laboratory values fall outside the UMHS normal ranges and are considered clinically significant will be required to have medical clearance from their primary care provider prior to participation. Potential subjects presenting with clinically insignificant laboratory abnormalities will not require medical clearance and will be considered for inclusion in the study
* Endocrine disorders/dysfunctions (i.e. Type I and II diabetes)
* Cancer - The explicit definition of cancer used to exclude patients is consistent with that described by the National Cancer Institute (NCI), National Institutes of Health. According to NCI, cancer is any disease in which abnormal cells divide without control and invade nearby tissues (invasive disease). These include carcinomas, sarcomas, leukemias, and lymphomas. Any patient with a history of these invasive diseases will be excluded from the study.
* Patients who currently use bisphosphonates or have a history of bisphosphonate use will be excluded from the trial
* HIV+
* Metabolic Bone Diseases- Patients with metabolic bone diseases such as Paget's disease, hypercalcemia, moderate to severe vitamin D3 abnormalities or any other metabolic bone disease including osteoporosis and osteoporotic fractures will be excluded
* Pregnant women- Female patients who are of childbearing potential are excluded except those who are using hormonal or barrier methods of birth control (oral or parenteral contraceptives, diaphragm plus spermicide, or condoms). Pregnancy status will be determined with a urine test and patients who are pregnant will be excluded
* Patients with acute sinusitis, or presenting any sinus pathology that would contraindicate sinus augmentation
* Patients with congenital or metabolic bone disorders
* Current smokers (have smoked within 6 mos. of study onset)
* Subjects with congenital, or co-morbid conditions that would affect the study outcome or interpretation of study results will be excluded
* Individuals who have a BMI outside normal limits that deems them overweight (BMI >25) will be excluded due to potential difficulties in locating appropriate surgical entry of the iliac crest during the bone marrow aspiration procedure
* Long term (>2 weeks) use of antibiotics in the past 3 months
* Periodontally unstable subjects
* Subjects having any extractions in the possible treatment area in the past 3 months
* Subjects that are edentulous

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Giannobile, DDS, DMedSc, Principal Investigator — University of Michigan
Locations (1):
- Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Albrektsson T, Branemark PI, Hansson HA, Lindstrom J. Osseointegrated titanium implants. Requirements for ensuring a long-lasting, direct bone-to-implant anchorage in man. Acta Orthop Scand. 1981;52(2):155-70. doi: 10.3109/17453678108991776. PMID 7246093
- [Background] Amler MH. The time sequence of tissue regeneration in human extraction wounds. Oral Surg Oral Med Oral Pathol. 1969 Mar;27(3):309-18. doi: 10.1016/0030-4220(69)90357-0. No abstract available. PMID 5251474
- [Background] Colter DC, Class R, DiGirolamo CM, Prockop DJ. Rapid expansion of recycling stem cells in cultures of plastic-adherent cells from human bone marrow. Proc Natl Acad Sci U S A. 2000 Mar 28;97(7):3213-8. doi: 10.1073/pnas.97.7.3213. PMID 10725391
- [Background] Krebsbach PH, Kuznetsov SA, Bianco P, Robey PG. Bone marrow stromal cells: characterization and clinical application. Crit Rev Oral Biol Med. 1999;10(2):165-81. doi: 10.1177/10454411990100020401. PMID 10759420
- [Background] Kaigler D, Mooney D. Tissue engineering's impact on dentistry. J Dent Educ. 2001 May;65(5):456-62. PMID 11425250
- [Background] Mankani MH, Kuznetsov SA, Wolfe RM, Marshall GW, Robey PG. In vivo bone formation by human bone marrow stromal cells: reconstruction of the mouse calvarium and mandible. Stem Cells. 2006 Sep;24(9):2140-9. doi: 10.1634/stemcells.2005-0567. Epub 2006 Jun 8. PMID 16763200
- [Background] Marei MK, Nouh SR, Saad MM, Ismail NS. Preservation and regeneration of alveolar bone by tissue-engineered implants. Tissue Eng. 2005 May-Jun;11(5-6):751-67. doi: 10.1089/ten.2005.11.751. PMID 15998216
- [Background] Nevins M, Giannobile WV, McGuire MK, Kao RT, Mellonig JT, Hinrichs JE, McAllister BS, Murphy KS, McClain PK, Nevins ML, Paquette DW, Han TJ, Reddy MS, Lavin PT, Genco RJ, Lynch SE. Platelet-derived growth factor stimulates bone fill and rate of attachment level gain: results of a large multicenter randomized controlled trial. J Periodontol. 2005 Dec;76(12):2205-15. doi: 10.1902/jop.2005.76.12.2205. PMID 16332231
- [Background] Atwood DA, Coy WA. Clinical, cephalometric, and densitometric study of reduction of residual ridges. J Prosthet Dent. 1971 Sep;26(3):280-95. doi: 10.1016/0022-3913(71)90070-9. No abstract available. PMID 5284182
- [Background] Evian CI, Rosenberg ES, Coslet JG, Corn H. The osteogenic activity of bone removed from healing extraction sockets in humans. J Periodontol. 1982 Feb;53(2):81-5. doi: 10.1902/jop.1982.53.2.81. PMID 6950085
- [Background] Friedenstein AJ, Ivanov-Smolenski AA, Chajlakjan RK, Gorskaya UF, Kuralesova AI, Latzinik NW, Gerasimow UW. Origin of bone marrow stromal mechanocytes in radiochimeras and heterotopic transplants. Exp Hematol. 1978 May;6(5):440-4. PMID 350596
- [Result] Kaigler D, Avila-Ortiz G, Travan S, Taut AD, Padial-Molina M, Rudek I, Wang F, Lanis A, Giannobile WV. Bone Engineering of Maxillary Sinus Bone Deficiencies Using Enriched CD90+ Stem Cell Therapy: A Randomized Clinical Trial. J Bone Miner Res. 2015 Jul;30(7):1206-16. doi: 10.1002/jbmr.2464. PMID 25652112

RESULTS

PARTICIPANT FLOW:
Groups:
- Sinus Lift Plus Dental Implant: Transalveolar sinus augmentation will be performed. After 4 months dental implants will be delivered only if primary stability can be achieved.
  Intervention (Procedure/Surgery): Sinus lift augmentation and dental implant transalveolar sinus augmentation will be performed. After 4 months, dental implants will be delivered only if primary stability can be achieved.
  Biological/Vaccine: N/A; only sinus augmentation and dental implant
  Sinus lift augmentation and dental implant: transalveolar sinus augmentation will be performed. After 4 months, dental implants will be delivered only if primary stability can be achieved.
- Sinus Lift Plus BRCs and Dental Implant: transalveolar sinus augmentation will be performed. A unit dose of BRC (10 ml) will be mixed with a commercially available β-TCP (Cerasorb), which will be used as a carrier to deliver the cells.
  Intervention (Procedure/Surgery): Sinus lift augmentation and dental implant transalveolar sinus augmentation will be performed. After 4 months, dental implants will be delivered only if primary stability can be achieved.
  Biological/Vaccine: Aastrom BRCs, sinus augmentation, BRC application, dental implant
  Aastrom BRCs: sinus augmentation, BRC application, dental implant
Period: Overall Study
Arm/Group | Sinus Lift Plus Dental Implant | Sinus Lift Plus BRCs and Dental Implant
Started | 13 | 13
Completed | 11 | 13
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sinus Lift Plus Dental Implant | Sinus Lift Plus BRCs and Dental Implant | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Customized [Number; unit: participants]
  >20 and <70 | 13 | 13 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density of Bone Core
Description: Bone mineral density of bone core was measured by histological and µCT analyses
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: mg/mm^3
Arm/Group | Sinus Lift Plus Dental Implant | Sinus Lift Plus BRCs and Dental Implant
Number analyzed (Participants) | 11 | 13
mg/mm^3 | .79 (.05) | .78 (.02)

2. Secondary Outcome: Change in Linear Radiographic Bone Height
Description: Change in linear radiographic bone heights were measured before and after bone graft reconstruction
Time Frame: Screening and 1 week post-op from baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Sinus Lift Plus Dental Implant | Sinus Lift Plus BRCs and Dental Implant
Number analyzed (Participants) | 11 | 13
mm | 12.8 (2.8) | 12.2 (3.3)

3. Primary Outcome: Bone Volume Fraction of Bone Core
Description: Bone volume fraction of bone core histological and µCT analyses
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sinus Lift Plus Dental Implant | Sinus Lift Plus BRCs and Dental Implant
Number analyzed (Participants) | 11 | 13
ratio | .43 (8.1) | .49 (7.2)

4. Secondary Outcome: Change in Sinus Bone Volume
Description: CBCT was used to evaluated 3-D changes in the bone volume within the treated areas of the sinus cavity
Time Frame: Pre-baseline and within 2 weeks of 4 Month visit
Measure: Mean (Standard Deviation); unit: cm3
Arm/Group | Sinus Lift Plus Dental Implant | Sinus Lift Plus BRCs and Dental Implant
Number analyzed (Participants) | 11 | 13
cm3 | 2.1 (.9) | 1.8 (1.0)

5. Secondary Outcome: Final Bone Volume: Initial Graft Volume Ratio
Description: Bone volume fraction of bone core histological and µCT analyses
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sinus Lift Plus Dental Implant | Sinus Lift Plus BRCs and Dental Implant
Number analyzed (Participants) | 11 | 13
ratio | .64 (.2) | .51 (.3)

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Sinus Lift Plus Dental Implant | Sinus Lift Plus BRCs and Dental Implant
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/13
Other Adverse Events (participants affected / at risk) | 9/13 | 9/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sinus Lift Plus Dental Implant (N=13) | Sinus Lift Plus BRCs and Dental Implant (N=13)
Sinus (Infections and infestations) | 0 (0) | 1 (13)
Surgery (Surgical and medical procedures) | 1 (13) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sinus Lift Plus Dental Implant (N=13) | Sinus Lift Plus BRCs and Dental Implant (N=13)
Lesion (General disorders) | 1 (1) | 0 (0)
Bleeding (General disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Soft Tissue Opening (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Broken Tooth (General disorders) | 2 (2) | 0 (0)
Suture Loss (General disorders) | 0 (0) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Shingles (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain and Swelling (General disorders) | 0 (0) | 2 (2)
Flap Mobility (General disorders) | 1 (1) | 0 (0)
Sore Throat (General disorders) | 0 (0) | 1 (1)
Non-restoreable Tooth (General disorders) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Headaches (General disorders) | 0 (0) | 1 (1)
Oral Ulcer (General disorders) | 1 (1) | 0 (0)
Tingling (General disorders) | 0 (0) | 1 (1)
Lack of Bone (General disorders) | 1 (1) | 1 (1)
Rash (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1)
Discomfort (General disorders) | 0 (0) | 1 (1)
Prosthesis Came Off (General disorders) | 6 (6) | 2 (2)
Swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sensitivity (General disorders) | 0 (0) | 1 (1)
Bleeding (General disorders) | 0 (0) | 1 (1)
Tenderness (General disorders) | 0 (0) | 1 (1)
Ovarian Ulcer Rupture (General disorders) | 1 (1) | 0 (0)
Exostosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Perforations (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No